CLINICAL TRIAL: NCT06541860
Title: Salvage Regimens in Multiple Myeloma Patients Double Refractory to Lenalidomide and MoAbs: Evidence From Real World Experience
Brief Title: DAratumumab and REvlimid REfractory MM
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: DARE-MM
Record Dates: First submitted 2024-04-09; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective and prospective multicenter observational study on patients with relapsed and refractory multiple myeloma after anti-CD38 MoAb therapy and IMIDS treated with onlabel regimens.

ELIGIBILITY:
Inclusion Criteria:

Phase I

* Patients with RRMM after therapy with anti-CD38 MoAb plus IMIDS started on therapy with PVD scheme
* Patients aged ≥ 18 years
* Patients able to understand and voluntarily sign an informed consent and be willing to consent to the review of clinical data

Phase II

* Patients with RRMM after first-line therapy with anti-CD38 MoAb plus IMIDS started on therapy with on-label schemes
* Patients aged ≥ 18 years
* Patients able to understand and voluntarily sign an informed consent and be willing to consent to the review of clinical data

Exclusion Criteria:

* Patients not willing to consent to review of clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed and refractory multiple myeloma after anti-CD38 MoAb therapy and IMIDS treated with onlabel regimens.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2028-02-21 (Estimated); Study Completion 2028-08-21 (Estimated)

PRIMARY OUTCOMES:
To explore the efficacy and tolerability of different combinations, particularly the PVD regimen, in the emerging context of RRMM after anti-CD38 MoAb plus IMIDS therapy. | 2 years
  Phase I - Retrospective study The primary objective is to estimate 2-year progression-free survival (PFS) of PVd when used in RRMM after anti-CD38 MoAb and IMIDS
  Phase II - Prospective study The primary objective is to estimate the 2-year progression-free survival (PFS) of the on-label combinations in patients with relapsed RRMM after first-line therapy with anti-CD38 MoAb plus IMIDS

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Matteo Pavia, Pavia, PV, Italy